CLINICAL TRIAL: NCT06554808
Title: Impact of Comorbidity on the Association Between Socioeconomic Factors and Long-term Mortality of Intensive Care Patients
Brief Title: Socioeconomic Factors and Mortality in the Intensive Care Population
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Anna Aronsson, PhD student, Uppsala University
Other Study IDs: UU Intensive Care
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Socio-economic Status; Comorbidity
Keywords: Critical care; Intensive care; Mortality; Socio-economic status; Comorbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Income: 1. 0-9999 Euros
  2. 10 000-29 999 Euros
  3. 30 000-49 999 Euros
  4. > 50 000 Euros
- Educational level: 1. Low - compulsory school (9 years)
  2. Medium - upper secondary school (additional 2-4 years)
  3. High - included education beyond that level (university)

SUMMARY:
It is important to find out how much of the socioeconomic factors´ impact on mortality on ICU patient´s can be explained by the presence of comorbidity. The aim of this study is to clarify the impact of socioeconomic factors on mortality and how much of this effect are due to comorbidity in the intensive care population.

DETAILED DESCRIPTION:
The first ICU admissions of patients aged 30 years and older, registered in the Swedish Intensive Care Registry (SIR) from 2009 to 2012 were included. SIR was linked to the National Patient Register, Statistics Sweden and the Cause of Death Register using unique person identity numbers. Educational level and disposable income was reported in the year preceding the admission to intensive care to not be affected by the current illness.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Swedish Intensive Care Registry (SIR) from 2009 to 2012.
* The first ICU admission
* Patients aged 30 years and older

Exclusion Criteria:

* Missing registration of educational level
* Missing registration of income

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first ICU admissions of patients aged 30 years and older, registered in the Swedish Intensive Care Registry (SIR) from 2009 to 2012.
Sampling Method: Non-Probability Sample
Enrollment: 101745 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | january 1, 2009 til december 31, 2016
  Mortality

IPD SHARING:
Plan to Share IPD: No
It is a register-based study where all the data are deidentified.